CLINICAL TRIAL: NCT04849546
Title: Assessment of the Physical and Mental Health of Private and Public Care Facilities Personnel in the Brestois Sector Following the First Peak of the Covid-19 Outbreak
Brief Title: Staff Physical and Mental Health Assessment in the Aftermath of the First Peak of the Covid-19 Outbreak
Acronym: SAMAF
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: SAMAF - 29BRC21.0125
Record Dates: First submitted 2021-04-15; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-02

CONDITIONS: Occupational Stress
Keywords: healtcare worker; COVID 19
MeSH Terms: conditions — Occupational Stress; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objectives: This study compare the mental health impact and psychosocial perception of healthcare workers and non healthcare workers in hospital after the first peak of COVID-19 outbreak in France.

Methods: The validated SATIN questionnaire with specific scoring was used to collect data on health and psychosocial factors. A self-administered online questionnaire was send to all workers of the hospital in June 2020. A multinomial regression model was created to assess differences and risk factors in outcomes between healthcare workers and non healthcare workers. Variables were adjusted for age, sexe, frontline workplaces and experience at hospital.

DETAILED DESCRIPTION:
The survey was conducted between 01 th of July and 31th of August 2020 and involved all workers employed in a teaching hospital in France. The total number of workers was 7299.

The Inclusion criteria were as follows: working in the hospital since more than one year, adults over than 18 years, acceptance.

Questionnaire After SATIN questionnaire authors allowing, we created a specific questionnaire with all original questions and some additional on workplaces and demographics' data. In first question, participants must check that they met inclusion criteria and accept to be included in this survey. An open question was available at the end for remarks.

86 questions in 6 parts: 1. Personnel and Professional Identification (10 questions) 2. Health reports (16 questions) 3. Work strain and capacities (8 questions) 4. Working environment (39 questions) 5. Work assessment (4 questions) 6. Supplementary questions for occupational physician (9 questions) Each question had five possible answers and each answer is linked to a specific score. Mean of scores were calculated in each part of the questionnaire: health reports (physical health, psychic health, physical symptoms, psycho-somatic symptoms, and stress), work strain and ability, working environment (physical environment, activity, framework of activities and organizational context), self-assessed work conditions in their entirety. The scores of each part were interpreted as follows: <2.5 poor health or negative perception, 2.5-3.5 mild health or perception, > 3.5 good health or positive perception. Global health and general workplace environment self-evaluation were scored in a second time with respectively health reports and working environment scores.

Demographic data were self-reported by the participants including occupation, sexe (male/female), age (<34, 35-44, 45-54, >55 years), time at workplace (<5, 6-15, 16-26,>26 years), shift work or night work (never, rarely, regularly, often/very often).

Statistical analyses. Data analysis was performed using R software (R Foundation for Statistical Computing, Vienna, Austria). The results for continuous variables were shown as medians with Interquartile range (IQRs). The ranked data, which were ranked from each part of the questionnaire, are presented as numbers and percentages. Participants were divided into three groups according to the previously reported questionnaire cut-off (<2.5; 2.5-3.5; > 3.5). Doctor, nurse, medical student, nurse assistant, midwife, paramedics, physiotherapist and radiographer were included in the subgroup "health care worker", other participants were included in the subgroup "non healthcare worker". We also made an analysis by subgroup of workers if they regularly or not worked in a COVID 19 dedicated sector. A multinomial logistic regression analysis was performed and the associations between risk factors and outcomes are presented as Odds Ratio (ORs) and 95% Confidence Intervals (Cis), after adjustment for cofounders including, gender, age, years at workplace. The significant level was set at p= 0.05.

ELIGIBILITY:
Inclusion Criteria:

* working in Brest teaching hospital or brest health clinic more than one year and aged> 18

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all workers from brest teaching hospital and private health clinic in Brest
Sampling Method: Non-Probability Sample
Enrollment: 1491 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
global health | july-august 2020
  Questionnaire on global health assessment with physical and psychological healt assessment and well being.

SECONDARY OUTCOMES:
psychosocial factors | july- august 2020
  validated questionnaire on psychosocial factors

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, Brittany Region, France